CLINICAL TRIAL: NCT06832098
Title: The New Zealand Quit Vaping Trial: Combination Nicotine Replacement Therapy Versus Nicotine Reduction.
Brief Title: Nicotine Patch Plus Nicotine Mouth Spray Versus Nicotine Reduction for Vaping Cessation
Acronym: EQUIT3
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Auckland, New Zealand (Other)
Collaborators: University College, London (Other); Medical University of South Carolina (Other); Flinders University (Other)
Responsible Party: Principal Investigator, George Laking, Associate Professor, University of Auckland, New Zealand
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U1111-1298-1142
Record Dates: First submitted 2025-02-04; First posted 2025-02-18 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Vaping Cessation
Keywords: Nicotine tapering; Pragmatic; Effectiveness; Vaping cessation; Nicotine Replacement Therapy; e-cigarette; nicotine mouth spray; nicotine patch
MeSH Terms: conditions — Vaping | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination NRT plus written behavioral support (Active Comparator): Participants allocated eight weeks of combination NRT (21mg patch plus 1mg mouth spray) will be advised to start using the patches daily, with the mouth spray used to relieve any 'breakthrough' cravings. Advice on reducing use of both products over the eight-week period will also be provided, following the manufacturers guidelines when these products are used for smoking cessation. Participants will also receive written behavioural support.
  Interventions: Combination Product: Nicotine patches plus nicotine mouth spray
- Nicotine Tapering Plan plus written behavioral support (Active Comparator): Participants allocated the eight-week nicotine tapering plan will be advised to follow the instructions provided. Participants will also receive written behavioural support.
  Interventions: Other: Nicotine Tapering Plan

INTERVENTIONS:
Combination Product: Nicotine patches plus nicotine mouth spray — Transdermal HABITROL® patches (21mg/24 hrs) plus NICORETTE® QUICKMIST mouth spray (1mg nicotine/spray dose)
  Other Names: HABITROL patches; NICORETTE QUICKMIST
  Arms: Combination NRT plus written behavioral support
Other: Nicotine Tapering Plan — Tapering plan based on their current e-juice nicotine concentration and frequency of vaping upon entry to the trial. Participants will use their own vapes and nicotine e-liquid.
  Arms: Nicotine Tapering Plan plus written behavioral support

SUMMARY:
This research focuses on maximizing the chances of successfully quitting vaping. A large, pragmatic community-based clinical trial is planned in New Zealand to build on existing evidence from previous vaping and smoking cessation research undertaken by the study team. The effectiveness of combination nicotine replacement therapy (NRT) compared to nicotine tapering on vaping abstinence has not yet been investigated, but both provide an opportunity to increase success with vaping cessation, especially when combined with written behavioural support to further boost quit rates.

The planned trial will test whether using combination NRT will help more New Zealanders to quit vaping long-term, compared with a vape nicotine tapering plan. Participants in both groups will also receive written vaping cessation behavioural support.

DETAILED DESCRIPTION:
Aim:

To evaluate the effectiveness, safety and acceptability of combination NRT plus behavioural support compared with vape nicotine tapering plus behavioural support, on six-month vaping abstinence.

Trial Design:

A single-blind, two-arm, pragmatic community-based randomised trial.

Eligibility criteria:

Eligible participants must live in New Zealand, vape nicotine at least weekly, used to smoke tobacco regularly but not in the past 6-months OR have never smoked tobacco, are aged ≥16 years, and have no contraindications to the study treatment. Participants must be motivated to quit-vaping in the next eight weeks, have access to the internet, and be able to provide consent. Participants must also have no treatment preference (i.e., they are happy to use whatever treatment they are allocated). Full details of inclusion and exclusion criteria are provided later in this trial registration.

Recruitment:

Participants will be recruited from throughout New Zealand, using multi-media advertising with targeted promotion to reach indigenous Māori, Pacific, low socio-economic groups, and people with disabilities, given their disproportionately higher prevalence of vaping. Advertisements will direct potential participants to a trial website where they can read the participant information sheet. A two step-consent process will be used. First, interested participants will be asked for on-line consent to complete an online screening questionnaire to determine their eligibility for the trial and verify their phone number. Second, eligible and interested participants will then provide online consent to enter the trial.

Baseline information:

Baseline data will then be collected via the online platform, and will include demographic data, body mass index, vaping history, vaping dependence, motivation to quit, signs and symptoms of nicotine withdrawal and urge to vape, smoking history, alcohol use, cannabis use, self-reported comorbidities, health-related quality of life, and concomitant medication. Full details on the baseline data are provided later in this trial registration. Once participants complete and submit the baseline form, they will be randomised to one of the two trial treatment groups and immediately notified of their allocated intervention.

Randomization:

Participants will be assigned a unique registration number allocated by a central computer, following details submitted via the website. Eligible participants will be randomised via computer (1:1 ratio) to one of two trial groups using stratified block randomisation (using varying block sizes), and stratified by ethnicity (Māori, non-Māori) and smoking status (never smoked, used to smoke). The randomisation sequence will be generated by the trial statistician, and centrally managed and concealed until the point of randomisation.

Blinding:

This is a single-blind trial as participants will be aware of the intervention to which they have been allocated, and data collection by the trial research assistants will include questions specific to use of participants allocated treatment. Except for the trial statistician, the trial steering committee members will remain blinded to treatment allocation until analyses are complete. The statistical analysis plan will be finalised and uploaded to the trial registry prior to the first participant being randomised.

Interventions:

Participants will be randomised to eight weeks of: 1) combination NRT (21mg patch plus 1mg mouth spray) or 2) a written vape nicotine tapering programme. Tapering will be based on the participants current e-juice nicotine concentration and frequency of vaping upon entry to the trial. Participants will use their own vapes and nicotine e-liquid. All participants will also receive written behavioural support which will focus on building self-efficacy and relapse prevention. All interventions will be couriered to participants immediately after randomization, at no cost to participants. The courier company will notify the study center immediately after the courier pack has been delivered, which will trigger the scheduling of the 'end of treatment' call (i.e., eight weeks after treatment delivery).

Follow-up:

Participants will be asked to begin their treatment the day after they receive their courier pack. Participants will be advised to continue with their allocated treatment, irrespective of any lapses back to vaping (or smoking), with the aim to be vape-free by the end of eight weeks (the designated quit date and end of treatment). All follow-up calls will be anchored to end of treatment (i.e., eight weeks after treatment delivery), whether they started or completed treatment.

Outcome data:

The primary outcome is being vape-free and tobacco-free, defined as self-reported continuous abstinence from vaping at six-months post-end of treatment. Specifically, self-report of no device use (defined as not vaping more than five vaping sessions since end of treatment), and no use of any tobacco products (defined as not smoking more than five cigarettes since end of treatment and no use of any other tobacco products since end of treatment), but individuals may or may not be using NRT. The primary outcome is partially validated. There is no vaping-specific biomarker available, so verification of 'vape-free' status can't be validated. However, tobacco-free status will be verified using exhaled carbon-monoxide (CO) measurement with a Bedfont Smokerlyzer (≤5 ppm signifying abstinence). Outcomes collected at end of treatment, then one-, three-, and six-months post end of treatment include other cessation outcomes, lapse/relapse to vaping, relapse to smoking in people who used to smoke, treatment adherence and compliance, other vaping support, signs and symptoms of nicotine withdrawal and urge to vape, cross-over, acceptability, recommendation of treatment to others, continuation of treatment, cannabis and alcohol use (six months only), change in body mass index, change in health state, serious adverse events, health-related quality of life, cost outcomes, concomitant medication, and participant experience in the trial. Full details on the outcome data are provided later in this registration.

Trial power:

A total of 774 participants (387 per group) will provide 90% power at p=0.05 to detect an absolute difference of 11% in self-reported six-month continuous abstinence rates (Vape-free and tobacco-free) between the combination NRT plus behavioural support group and the vape nicotine tapering plus behavioural support group. We have assumed that the self-reported six-month continuous abstinence vaping quit rates (vape-free and tobacco-free) for those in the NRT group will be 26%, compared to 15% in the nicotine tapering group. The sample size accounts for a 28% loss-to-follow-up at six months.

Statistical analysis:

All statistical analyses will be performed using SAS version 9.4 (SAS Institute Inc. Cary NC), and R. Data analyses will be specified a priori in a statistical analysis plan prepared by the trial statistician and posted on the trial registry prior to the first participant recruitment. No interim analyses will be undertaken. All analyses will be conducted for combination NRT plus behavioural support compared with the vape nicotine tapering plus behavioural support. The main analyses will be carried out on an intention-to-treat basis, with multiple imputation analysis performed to account for missing data using the fully conditional specification logistic regression method (data will be assumed to be missing at random).

ELIGIBILITY:
Inclusion Criteria:

* Live in New Zealand.
* Vape nicotine at least weekly (one or more days out of the past seven days).
* Used to smoke (i.e. they have smoked tobacco regularly but not at all in the past six months) or have never smoked (i.e., they have never been a regular user of smoked tobacco, defined as less than 100 cigarettes in their lifetime).
* Are aged ≥16 years.
* Are motivated to quit vaping in the next eight weeks.
* Are able to provide consent.
* Have access to the internet via a computer or smart phone.
* Are a registered patient at a New Zealand medical facility.

Exclusion Criteria:

* They have another person in their household currently enrolled in the study.
* They smoke tobacco currently or were a recent regular user of tobacco.
* They are enrolled in another vaping cessation programme/trial.
* They self-report having had a serious cardiovascular event, or hospitalisation for a cardiovascular complaint, in the previous four weeks (e.g. stroke, myocardial infarction, unstable angina, cardiac arrhythmia, coronary artery bypass graft and angioplasty).
* They self-report uncontrolled hypertension.
* They have a strong preference to use/not use NRT or nicotine tapering.
* They are current users of smoking cessation pharmacotherapy (e.g. NRT, varenicline, cytisine, nortriptyline [including if it is used for a different indication], and amitriptyline [as it converts to nortriptyline].
* They are currently enrolled in another vaping cessation programme/trial.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 774 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Vape-free and tobacco-free: self-reported continuous abstinence from vaping at six-months post-end of treatment | Six months post-end of treatment
  Self-report of no device use (defined as not more than five vaping sessions since end of treatment), and self-report of not smoking (defined as no use of any tobacco, but individuals may or may not be using NRT. The tobacco-free status will be verified using exhaled carbon-monoxide (CO) measurement with a Bedfont Smokerlyzer (≤5 ppm signifying abstinence).

SECONDARY OUTCOMES:
Age | Baseline
  Date of birth will be recorded to enable the age at baseline to be reported for each treatment group (presented as a mean, and associated standard deviation, or median and inter-quartile range).
Gender | Baseline
  Gender will be reported as counts and proportions of male, female, and gender diverse at baseline, for each treatment group.
Ethnicity (self-reported) | Baseline
  Ethnicity will be reported as counts and proportions of Maori, Pacific or Other, for each treatment group.
Education | Baseline
  Education level will be reported as counts and proportions of participants with "less than 12 years of attending school" or "12 or more years of attending school" or "prefer not to answer", for each treatment group.
Number of years of continuous vaping | Baseline
  Participants will be asked how many years they have been vaping continuously, with results presented as a mean with the associated standard deviation (or median and interquartile range) for each treatment group.
Age started vaping | Baseline
  The age participants started vaping will be reported, with results presented as a mean and associated standard deviation for each treatment group, or median and interquartile range.
Previous quit attempts | Baseline
  Participants will be asked if they have tried to quit vaping before (Yes/No), with data reported as counts and proportions for each treatment group.
Number of serious quit attempts | Baseline
  [If outcome 8 is answered YES] Participants will be asked about the number of serious quit attempts they have made (i.e., 0, 1, 2, 3, 4, 5 or more), with data presented as counts and proportions for each treatment group. "Serious attempt" is defined as they decided they would try to make sure they never vaped again.
Longest time being vape-free in the last 12 months | Baseline
  [If outcome 9 is answered 1 or more] Participants will be asked about how long (in days) they managed to stop vaping in the last 12 months. This question is a free text field. Data will be grouped and reported as counts and proportions for each treatment group.
Methods used to stop vaping during the last serious attempt | Baseline
  [If outcome 9 is answered 1 or more] Participants will be asked what methods they used to stop vaping, during their most recent quit attempt. Methods will include: Nothing, Support from former and/or current vapers, Support from my friends and/or family, Support from my workplace, Support from Quitline or another smoking cessation service, I tried reducing the strength of the nicotine over time, Nicotine patches, Nicotine gum, Nicotine lozenges, Nicotine mouth spray, Champix (varenicline), Cytisine, an app (asked for app name), Prayer, Something else (free text option). Multiple options can be chosen. Results will be reported as counts and proportions for each treatment group.
Vape type | Baseline, eight weeks (i.e., end of treatment), then at one-, three-, and six-months post end of treatment
  Participants will be asked what type of vape they are currently using. Options are a disposable device; a rechargeable device with pods; a rechargeable device with a refillable tank; a modifiable device, Other (free text option). Data presented as counts and proportions for each treatment group.
Use of a nicotine salt | Baseline, eight weeks (i.e., end of treatment), then at one-, three-, and six-months post end of treatment in those still vaping
  Participants will be asked if they vape a nicotine salt. (Yes, No, Sometimes, Don't know), with data presented as counts and proportions for each treatment group.
Strength of nicotine used | Baseline, eight weeks (i.e., end of treatment), then at one-, three-, and six-months post end of treatment in those still vaping nicotine
  Participants will be asked what nicotine strengths they currently use (0mg or 0.0%; 1-3mg or 0.1-0.3%; 4-12mg or 0.4-1.2%; 13-28.5mg or 1.3-2.85%; More than 28.5mg or 2.85%; There is nicotine in the vape, but I don't know the strength; Don't know), with data presented as counts and proportions for each treatment group. Multiple options are permitted.
Vape flavor | Baseline, eight weeks (i.e., end of treatment), then at one-, three-, and six-months post end of treatment in those still vaping nicotine
  Participants will be asked what flavors they currently vape (Mint/Menthol; Tobacco; Fruit; Combination such as mint + fruit; Other [free text]). Multiple options are permitted. Results will be presented as counts and proportions for each treatment group.
Frequency of vaping in the last seven days | Baseline
  Participants will be asked how often they vaped in the last seven days, with answer options of: Everyday; Six of the 7 days; Five of the 7 days; Four of the 7 days; Three of the 7 days; Two of the seven days; and On one day only. Data will be presented as counts and proportions for each treatment group.
Frequency of vaping on the days they vaped in the last seven days (Baseline) | Baseline
  Participants will be asked how often they vaped, on the days they vaped in the last seven days (i.e., how many times they vaped on and off for 5 minutes or more). Free text field. Data will be grouped and presented as counts and proportions.
Money spent on vaping in last 7 days | Baseline, eight weeks (i.e., end of treatment), then at one-, three-, and six-months post end of treatment
  Participants will be asked about how much money they spend on vaping during the week (on average), with answer options of $0-10; $11-20; $21-30; $31-40; $41-50; more than $50. Counts and proportions will be presented for each treatment group.
Vaping of other substances | Baseline, eight weeks (i.e., end of treatment), then at one-, three-, and six-months post end of treatment
  Participants will be asked if they have vaped substances other than nicotine, reported as counts and percentages responding 'Yes' or 'No', for each treatment group.
Name of other substances vaped | Baseline, eight weeks (i.e., end of treatment), then at one-, three-, and six-months post end of treatment
  [Asked of those who answer YES to outcome 19] Participants will be asked what other substances they have vaped. This is a free text field. Results will be grouped by substance and reported as counts and percentages for each treatment group.
Vaping dependence | Baseline
  Vaping dependence will be determined using the validated 4-item e-cigarette dependence scale, with each item scored using a Likert scale of 0 "never" to 4 "almost always". Higher scores indicate higher levels of dependence, with scores ranging from 0 to 16). Results will be presented as a mean (with the associated standard deviation) for each treatment group.
Motivation to quit vaping | Baseline
  Motivation to quit vaping, measured using a five-point Likert Scale, where 1=not very motivated and 5=very motivated. Results will be presented as a mean with the associated standard deviation (or median and interquartile range) for each treatment group.
Self-rated chances of giving up vaping for good this time | Baseline
  Self-rated chances of giving up vaping for good this time, measured using a five-point Likert Scale, where 1=extremely low and 5=extremely high. Results will be presented as a mean with the associated standard deviation (or median and interquartile range) for each treatment group.
Live with people who smoke tobacco | Baseline
  Participants will be asked if they live with people who smoke (Yes; No; Sometimes). Results will be presented as counts and proportions for each treatment group.
Lives with people who vape | Baseline
  Participants will be asked if they live with people who vape (Yes; No; Sometimes). Results will be presented as counts and proportions for each treatment group.
Smoking history | Baseline
  Participants will be asked if they have ever regularly smoked tobacco in cigarettes, roll-your-owns, cigars, cigarillos, pipes, and/or shisha or water pipe. Answer options include: I have never smoked tobacco; I used to smoke tobacco, but don't now. Data will be reported as counts and proportions for each treatment group.
Frequency of smoking in those that smoked tobacco | Baseline
  [Asked of those who answered outcome 26 "I used to smoke tobacco, but don't now"]. Participants will be asked about how often they smoked, when they used to smoke. Answer options are: Everyday; not every day. Data will be reported as counts and proportions for each treatment group.
Age started smoking | Baseline
  [Asked of those who answered outcome 26 "I used to smoke tobacco, but don't now"]. Participants will be asked at what age they started smoking, with results presented as a mean with the associated standard deviation (or median and interquartile range) for each treatment group.
Number of years of continuous smoking | Baseline and six-months post end of treatment
  [Asked of those who answered outcome 26 "I used to smoke tobacco, but don't now"]. Participants will be asked how many years they smoked continuously, with results presented as a mean with the associated standard deviation (or median and interquartile range) for each treatment group.
Cannabis use | Baseline and six-months post end of treatment
  Participants will be asked how often they have used cannabis in the past six months (never, monthly or less, 2-4 times a month, 2-3 times a week, 4 or more times a week). This will be dichotomised to never used and have used cannabis in the past six months. Results will be presented as counts and proportions for each treatment group. Data will be reported as counts and proportions for each treatment group.
Change from baseline in alcohol use | Baseline and six-months post end of treatment
  Alcohol use will be measured using the three item Alcohol Use Disorders Identification Test (AUDIT-C). Item 1 asks "How often have you had a drink containing alcohol?" Item 2 asks with options of: Never (score=0); Monthly or less (score=1); 2-4 times per month (score=2); 2-3 times per week (score=3); 4 or more times a week (score=4). Item 2 asks "How many drinks do you usually have if you are drinking" with options of: 1 or 2 (score=0); 3 or 4 (score=1); 5 or 6 (score=2); 7 to 9 (score=3); 10 or more (score=4). Item 3 asks "How often have you had six or more drinks on one occasion?" with options of: Never (score=0); Less than monthly (score=1); Monthly (score=2); Weekly (score=3); Daily or almost daily (score=4). A total score ranges from 0 to 12. Higher scores indicate greater risk of alcohol dependence. Results will be presented as a mean (with the associated standard deviation) by gender each treatment group.
Change from baseline in body mass index | Baseline, eight weeks (i.e., end of treatment), then one-, three-, and six-months post end of treatment
  Self-reported height (m) and weight (kg) will be measured at baseline and combined to determine baseline body mass index (kg/m2). Self-reported weight (kg) will be asked at baseline, end of treatment, then at one, three, and six-months post end of treatment. Body mass index will be calculated for each timepoint to determine change in body mass index from baseline in those participants that quit vaping at these timepoints, compared to those that did not quit vaping.
History of mental health concerns | Baseline
  Participants will be asked if they have ever received medical treatment in the past for any mental health concerns: depression; schizophrenia or related disorder; anxiety; another mental health concern (free text), none of the above. Data will be reported as counts and proportions for each treatment group.
Current mental health concerns | Baseline
  Participants will be asked if they are currently receiving medical treatment for any mental health concerns, with answer options of: depression; schizophrenia or related disorder; anxiety; another mental health concern (free text), none of the above. Data will be reported as counts and proportions for each treatment group.
Change from baseline in severity of mental health concerns, in those participants with mental health concerns. | Eight weeks (i.e., end of treatment), then one-, three-, and six-months post end of treatment
  Participants who report at baseline that they are currently receiving treatment for any mental health concerns will be asked at follow-up whether their mental health symptoms have been: much worse; a bit worse; about the same; a bit better; or much better since starting the study. Data will be reported as counts and proportions for each treatment group.
Asthma | Baseline
  Participants will be asked at baseline if they have asthma (self-reported: Yes/No). Data will be reported as counts and proportions for each treatment group.
Change from baseline in asthma severity, in those participants with asthma | Baseline, eight weeks (i.e., end of treatment), then one-, three-, and six-months post end of treatment
  Participants who report at baseline that they have asthma will be asked at all follow-up time-points whether their asthma has been: much worse; a bit worse; about the same; a bit better; or much better since starting the study. Data will be reported as counts and proportions for each treatment group.
Chronic Obstructive Pulmonary Disease (COPD) | Baseline
  Participants will be asked at baseline if have COPD (self-reported: Yes/No). Data will be reported as counts and proportions for each treatment group.
Change from baseline in severity of COPD, in those participants with COPD. | Baseline, eight weeks (i.e., end of treatment), then one-, three-, and six-months post end of treatment
  Participants who report that they do have COPD will be asked at all follow-up time points whether their COPD has been: much worse; a bit worse; about the same; a bit better; or much better since starting the study. Data will be reported as counts and proportions for each treatment group.
Chronic pain | Baseline
  Participants will be asked at baseline if have chronic pain (self-reported: Yes/No). Data will be reported as counts and proportions for each treatment group.
Change from baseline in severity of chronic pain, in those participants with chronic pain. | Baseline, eight weeks (i.e., end of treatment), then one-, three-, and six-months post end of treatment
  Participants who report that they do have chronic pain at baseline will be asked at all follow-up points whether their chronic pain has been: much worse; a bit worse; about the same; a bit better; or much better since starting the study. Data will be reported as counts and proportions for each treatment group.
Frequency of coughing | Baseline
  Self-reported frequency of coughing will be measured at baseline (How often do you cough in your normal everyday life)? Response options are: Not at all; A little of the time; Some of the time; A lot of the time; All of the time). Data will be reported as counts and proportions for each treatment group.
Change from baseline in frequency of coughing | Baseline, eight weeks (i.e., end of treatment), then one-, three-, and six-months post end of treatment
  Self-reported frequency of coughing will be measured at each follow-up time point (How often do you cough in your normal everyday life)? Response options are: Not at all; A little of the time; Some of the time; A lot of the time; All of the time). Data will be reported as counts and proportions for each treatment group.
Frequency of shortness of breath | Baseline
  Self-reported frequency of shortness of breath will be measured at baseline (How often do you get short of breath? Response options are: Not at all; A little of the time; Some of the time; A lot of the time; All of the time). Data will be reported as counts and proportions for each treatment group.
Change from baseline in frequency in shortness of breath | Baseline, eight weeks (i.e., end of treatment), then one-, three-, and six-months post end of treatment
  Self-reported frequency of shortness of breath will be re-assessed at all follow-up time points (How often do you get short of breath? Response options are: Not at all; A little of the time; Some of the time; A lot of the time; All of the time). Data will be reported as counts and proportions for each treatment group.
Health-related quality of life (five domains) | Baseline
  Measured using the EQ-5D-5L - a standardized measure of health-related quality of life developed by the EuroQol Group. EQ-5D-5L is not an abbreviation. The EQ-5D-5L consists of five questions - each describe a different dimension of health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five levels: no problems, slight problems. moderate problems, severe problems, extreme problems (labelled 1-5). Answers will be valued (weighted to New Zealand population norms) and transformed into a utility score using a scoring algorithm and presented as a mean (with the associated standard deviation) for each treatment group.
Health-related quality of life (five domains) | Baseline, eight weeks (i.e., end of treatment), then one-, three-, and six-months post end of treatment
  Measured using the EQ-5D-5L - a standardized measure of health-related quality of life developed by the EuroQol Group. EQ-5D-5L is not an abbreviation. The EQ-5D-5L consists of five questions - each describe a different dimension of health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five levels: no problems, slight problems. moderate problems, severe problems, extreme problems (labelled 1-5). Answers will be valued (weighted to New Zealand population norms) and transformed into a utility score using a scoring algorithm and presented as a mean (with the associated standard deviation) for each treatment group.
Change in signs and symptoms of nicotine withdrawal in participants | Baseline, eight weeks (i.e., end of treatment), one-, three-, and six-months post end of treatment
  Measured using the Mood and Physical Symptoms Scale (MPSS) which consists of 5-point ratings of depressed mood, irritability, restlessness, hunger and difficulty concentrating. The MPSS score is calculated by summing all 5 items (scored 1-5: not at all, slightly, moderately, very, extremely) and has a range of 5 to 25, where higher scores indicate greater nicotine withdrawal. Scores will be presented as a mean with the associated standard deviation, for each treatment group.
Change in urge to vape | In last eight weeks (measured at end of treatment), and one-, three-, and six-months post end of treatment
  Measured using a 6-point rating of time spent with an urge to vape (scored 0-5: not at all, a little of the time, some of the time, a lot of the time, almost all of the time, all of the time), and the strength of these urges over the past week (scored 0-5: no urges, slight, moderate, strong, very strong, extremely strong). Participants who tick 'Not at all' for time spent with urges to vape, then skip to the next section of questions and don't answer the question on strength of urges. For these participants the strength of urges is set at 0, therefore, this question will then have values 0 to 5. The urge score is calculated by summing the two urges questions and has a range 0 to 10, where higher scores indicate greater urge to smoke. Scores will be presented as a mean with the associated standard deviation, for each treatment group
Vape-free and tobacco-free (self-reported continuous abstinence) | Eight weeks (i.e., end of treatment), then one-, three-, and six-months post end of treatment
  Defined as self-reported continuous abstinence from vaping since end of treatment (i.e., no more than five vaping sessions since end of treatment) and no tobacco use (i.e. not smoking more than five cigarettes and no use of any tobacco products since end of treatment) - but may or may not be using nicotine replacement therapy
Vape-free and tobacco-free (self-reported point prevalence abstinence) | In last eight weeks (measured at end of treatment), and one-, three-, and six-months post end of treatment
  Defined as self-reported 7-day point prevalence abstinence from vaping since end of treatment (i.e., no more than five vaping sessions in the last 7 days and no tobacco use in the last 7 days (not even a single puff/use), but may or may not be using nicotine replacement therapy.
Vape-free (self-reported continuous abstinence) | Eight weeks (i.e., end of treatment), then one-, three-, and six-months post end of treatment
  Defined as self-reported continuous abstinence from vaping since end of treatment (i.e., no more than five vaping sessions since end of treatment) - but may or may not be using tobacco and/or nicotine replacement therapy.
Vape-free (self-reported point prevalence abstinence) | One-, three-, and six-months post end of treatment
  Defined as self-reported 7-day point prevalence abstinence from vaping since end of treatment (i.e., no more than five vaping sessions in the last 7 days) - but may or may not be using tobacco and/or nicotine replacement therapy.
Nicotine-free (self-reported continuous abstinence) | One-, three-, and six-months post end of treatment
  Defined as self-reported continuous abstinence from nicotine since end of treatment, i.e., not vaping nicotine (not vaping nicotine more than five vaping sessions since end of treatment), not using tobacco ((not smoking more than five cigarettes and no use of any other tobacco products since end of treatment), and not using any nicotine replacement therapy since end of treatment.
Nicotine-free (verified continuous abstinence) | One-, three-, and six-months post end of treatment
  Verified six-month continuous abstinence from nicotine, defined as not vaping nicotine (not vaping nicotine more than five vaping sessions since end of treatment,), not using any tobacco products (not smoking more than five cigarettes and no use of any other tobacco products since end of treatment,), and not using any nicotine replacement therapy since the end of treatment. Abstinence will be verified using salivary cotinine (an established marker for nicotine from nicotine replacement therapy, vapes and tobacco) where a reading of ≤10 ng/ml signifies abstinence. Samples will be obtained from participants in the greater Auckland region who claim they are nicotine-free. sample results will be extrapolated to the full trial sample (Note: we do not have the funding to collect and test saliva samples from across all of New Zealand).
Nicotine-free (self-reported point prevalence abstinence) | One-, three-, and six-months post end of treatment
  Defined as self-reported 7-day point prevalence abstinence from nicotine since end of treatment, i.e., not vaping nicotine in the last 7 days, not using tobacco in the last 7 days (not even a single puff/use), and not using nicotine replacement therapy in the last 7 days.
Vaping (even a single puff) post end of treatment | One-, three-, and six-months post end of treatment
  Participants will be asked if they have vape (even a single puff) since the last contact post end of treatment, with answer options of: none, Yes a few puffs; Yes, 1 vaping session; Yes, 2 vaping sessions; Yes, 3 vaping sessions; Yes, 4 vaping sessions; Yes, 5 vaping sessions; Yes, more than 5 vaping sessions. A vaping cessation is defined as vaping on and off for 5 minutes or more. Data will be presented as counts and proportions for each treatment group.
Frequency of vaping in the last 7 days in those still vaping (post end of treatment) | One-, three-, and six-months post end of treatment
  Participants will be asked how often they vaped in the last seven days, with answer options of: no, not even a puff; yes, a few puffs; Yes, between 1 and 5 vaping sessions, yes, more than 5 vaping sessions. Data will be presented as counts and proportions for each treatment group.
Return to daily vaping (post end of treatment) | One-, three-, and six-months post end of treatment
  Participants will be asked if they have gone back to vaping daily (Yes or No). Data will be presented as counts and proportions for each treatment group.
Average vaping sessions per day, in those that are vaping everyday | One-, three-, and six-months post end of treatment
  [Those that respond Yes to Outcome 59]: Those that are vaping every day will be asked for the average number of vaping sessions per day [free text]. Data will be presented as means and standard deviations for each treatment group.
Time to first lapse back to vaping | One-, three-, and six-months post end of treatment
  Defined as time to first use of a vape since end of treatment, even a single puff.
Time to first relapse back to vaping | One-, three-, and six-months post end of treatment
  Defined as time to having more than 5 vaping sessions per day for 3 or more days in a row, since end of treatment.
Tobacco use in participants who have never smoked | Eight weeks (i.e., end of treatment), then one-, three-, and six-months post end of treatment
  Participants who have never smoked will be asked at each follow-up call whether they have smoked any tobacco since starting the trial (even just a puff). Answer options include: No, Yes - manufactured cigarettes, Yes - roll-your-own cigarettes, Yes- cigars, Yes - cigarillos, Yes - pipe, Yes - shisha / water pipe, Yes - other [free text field]. Multiple 'Yes' options can be chosen. Data will be reported as counts and proportions for each treatment group.
Frequency of smoking in participants who have never smoked (but have smoked tobacco since starting the trial) | Eight weeks (i.e., end of treatment), then one-, three-, and six-months post end of treatment
  Asked of those who answered 'Yes' to outcome 63. Participants will be asked how often they have smoked tobacco since starting the trial. Answer options are: daily; not every day, Just once or twice. Data will be reported as counts and proportions for each treatment group
Cigarettes smoked each day in participants who have never smoked (but currently smoke tobacco daily) | Eight weeks (i.e., end of treatment), then one-, three-, and six-months post end of treatment
  Asked of those who answered 'daily' to outcome 64. Participants will be asked about the number of cigarettes they smoke each day, with results presented as a mean (with the associated standard deviation) for each treatment group.
Cigarettes smoked per day (in participants who used to smoke, but have returned to smoking) | Eight weeks (i.e., end of treatment), then one-, three-, and six-months post end of treatment
  Number of cigarettes smoked per day, presented as summary statistics (mean, median, standard deviation, IQR)
Time to first lapse back to smoking (in participants who used to smoke) | One-, three-, and six-months post end of treatment
  Defined as time to first cigarette smoked since end of treatment, even a single puff.
Time to first relapse back to smoking (in participants who used to smoke) | One-, three-, and six-months post end of treatment
  Defined as time to smoking more than five cigarettes a day for three or more days in a row.
Number of self-reported serious adverse events | Eight weeks (i.e., end of treatment), then one-, three-, and six-months post end of treatment
  Only serious adverse events (SAEs) will be collected, given the well-known safety profile of NRT. Participants will be asked at each follow-up call about any new, unusual, unexpected serious adverse events during or since starting treatment, and whether they felt the event was related to treatment. SAEs will be classified as death, life threatening, hospitalization, persistent or sustained disability/incapacity, congenital abnormality/birth defect, or significant medical event. The likelihood of causality will be assessed using the World Health Organization Standardized Case Causality Assessment Tool (certain, probable/likely, possible, unlikely, conditional/unclassified, unassessable/unclassifiable). Data will be summarized as counts and percentages, according to treatment group.
Continuation of product use | Eight weeks (i.e., end of treatment), then one-, three-, and six-months post end of treatment
  Defined as continued use of the allocated treatment by participants after the end of the designed 8-week treatment period. Participants in the NRT group will also be asked if they used other forms of NRT, such as nicotine gum, lozenges, etc.
Use other vaping cessation support | Eight weeks (i.e., end of treatment)
  Participants will be asked about the use of other vaping cessation support, (i.e., support from former/current vapers; friends and/or family; work-place; Quitline or another smoking cessation service, own tapering plan; Nicotine patches; Nicotine gum; Nicotine lozenges; Nicotine mouth spray; Champix (varenicline); Cytisine; An app; Prayer; Complementary/alternative therapy or natural health product(s); Something else [free text]. Multiple answers options are permitted. Data will be reported as counts and proportions for each treatment group.
Participants recommendations regarding the allocated product | Eight weeks (i.e., end of treatment)
  Participants will be asked if they would recommend the allocated treatment to another person who vaped and wanted to quit (Answer options of: Yes; No]. People allocated the NRT will also have the answer options of "recommend mouth spray only' and "recommend nicotine patch only'. Data will be reported as counts and proportions for each treatment group.
Acceptability of the allocated intervention | Eight weeks (i.e., end of treatment)
  Participants will be asked for their views on the use of the allocated product(s) as a cessation aid, that is what participants liked or disliked about using the product(s): Answers will be provided as free text and summarized thematically.
Marginal cost per quitter | Eight weeks (i.e., end of treatment), then one-, three-, and six-months post end of treatment
  If the nicotine replacement therapy treatment is superior to the tapering plan, a cost-effectiveness analysis will be undertaken.
Treatment crossover | Eight weeks (i.e., end of treatment), then one-, three-, and six-months post end of treatment
  Participants in the nicotine reduction group will be asked whether they accessed and used nicotine patches and/or mouth spray during the trial, and if so, at what time during the trial and what product and nicotine strength they used. Participants in the nicotine reduction group will also be asked if they used other forms of NRT, such as nicotine gum, lozenges, etc, during the trial, with results reported as the counts and proportion at each time period.
Engagement with treatment | Eight weeks (i.e., end of treatment), then one-, three-, and six-months post end of treatment
  Participants will be asked about use of their allocated intervention. Engagement in the NRT group will be defined as use of their allocated interventions (patches and/or mouth spray) at least once during first two weeks (Yes/No). Engagement in the tapering group will be defined as reading and/or using the tapering plan at least once in the first two weeks (Yes/No).
Treatment use | Eight weeks (i.e., end of treatment)
  Participants allocated nicotine replacement therapy will be asked to provide a count of how much of the provided NRT they still have at end of treatment. Both groups will be asked about use of their allocated intervention at least once in the last 8 weeks (during the intervention period).

CONTACTS AND LOCATIONS:
Overall Officials: George Laking, PhD, MBChB, Principal Investigator — University of Auckland, New Zealand
Locations (1):
- School of Population Health, Faculty of Medical and Health Sciences, University of Auckland, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
This plan is currently being developed and will be made available soon. Please note that at least 25% of trial participants are likely to be Indigenous Māori. In New Zealand "indigenous data sovereignty recognizes that Māori data should be subject to Māori governance. Māori data sovereignty supports tribal sovereignty and the realization of Māori and Iwi aspirations." Requests to access trial data provided by Māori participants will be reviewed and considered by Dr George Laking (an indigenous Māori member of the trial steering committee).
Supporting Information: SAP
Time Frame: Data requests can be submitted starting nine months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Requests for access to individual participant data, or trial documents, will be considered where: 1) the request is from qualified researchers engaging in independent scientific research; 2) the proposed use aligns with public good purposes; 3) a research proposal and Statistical Analysis Plan are provided for review and approval; 4) the request does not conflict with other requests or planned use by members of the trial steering committee; and 5) the requestor is willing to sign a data access agreement. Please send all requests to the principal investigator.

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-02-21): https://cdn.clinicaltrials.gov/large-docs/98/NCT06832098/SAP_001.pdf